CLINICAL TRIAL: NCT02589392
Title: Effect of Cetaphil® Restoraderm® Moisturizer on Very Dry Skin in Children With a Controlled Atopic Dermatitis:a Randomised, Parallel Group Study
Brief Title: Cetaphil Restoraderm Effect on Young Children With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RD.03.SPR.29110
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moisturizer + Body wash (Experimental): Cetaphil® Restoraderm® moisturizer (2/day) + Cetaphil® Restoraderm® Skin body wash (1/day)
  Interventions: Other: Cetaphil® Restoraderm® moisturizer + Cetaphil® Restoraderm® body wash
- Body wash (Active Comparator): Cetaphil® Restoraderm® body wash (1/day)
  Interventions: Other: Cetaphil® Restoraderm® body wash

INTERVENTIONS:
Other: Cetaphil® Restoraderm® moisturizer + Cetaphil® Restoraderm® body wash
  Arms: Moisturizer + Body wash
Other: Cetaphil® Restoraderm® body wash
  Arms: Body wash

SUMMARY:
The purpose of this study is to evaluate the effect of Cetaphil® Restoraderm® skin restoring moisturizer in reducing the signs and symptoms of very dry atopic skin in young children. Subjects with atopic dermatitis (AD) in remission phase will be randomized to receive either Cetaphil® Restoraderm® skin restoring body wash only, or the same body wash in association with Cetaphil® Restoraderm® skin restoring moisturizer.

DETAILED DESCRIPTION:
Two groups randomized in a ratio of [1:1] for a 12-week period Five study evaluation were planned: at Baseline, week 2, Week 4, Week8 and Week12

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, aged 2 to 12 years inclusive
* Controlled mild to moderate atopic dermatitis with a Investigator Global Assessment score at 0 or 1, within one week after successful treatment with topical corticosteroid.

Exclusion Criteria:

* Subject presenting bacterial, viral, fungal or parasite skin infection
* Subject with ulcerated lesions, acne or rosacea
* Immunosuppression
* Subject with a wash-out period from baseline for topical treatment less than 8 days for Calcineurin inhibitor
* Subject with a wash-out period from baseline for topical treatment more than 8 days for corticosteroid
* Subject with a wash-out period from baseline for systemic treatment less than 8 days for anti-histamines, less than 4 weeks for immunomodulators

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- China (4):
  - Department of Dermatology /Shenzhen Children's hospital, Shenzhen, Guangdong
  - Hunan Children's Hospital, Hunan, Hunan
  - XinHua Hospital, Yangpu, Shanghai Municipality
  - Department of Dermatology /Beijing Children's Hospital, Beijing, XI Cheng
- Philippines (4):
  - Philippine General Hospital, Manila, Ermita
  - Asian Hospital and Medical Center, Manila, Muntinlupa City
  - St. Luke's Medical Center, City of Taguig, Taguig City
  - Jose R. Reyes Memorial Medical Center, Manila

REFERENCES:
- [Derived] Ma L, Li P, Tang J, Guo Y, Shen C, Chang J, Kerrouche N. Prolonging Time to Flare in Pediatric Atopic Dermatitis: A Randomized, Investigator-Blinded, Controlled, Multicenter Clinical Study of a Ceramide-Containing Moisturizer. Adv Ther. 2017 Dec;34(12):2601-2611. doi: 10.1007/s12325-017-0640-6. Epub 2017 Nov 16. PMID 29143926

RESULTS

PARTICIPANT FLOW:
Groups:
- Moisturizer + Body Wash: Cetaphil® Restoraderm® moisturizer (2/day) + Cetaphil® Restoraderm® Skin body wash (1/day)
  Cetaphil® Restoraderm® moisturizer + Cetaphil® Restoraderm® body wash
- Body Wash: Cetaphil® Restoraderm® body wash (1/day)
  Cetaphil® Restoraderm® body wash
Period: Overall Study
Arm/Group | Moisturizer + Body Wash | Body Wash
Started | 60 | 60
Completed | 54 | 54
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Sponsor decision to withdraw subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moisturizer + Body Wash | Body Wash | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (2.9) | 5.9 (2.9) | 5.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 23 | 27 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 60 | 58 | 118
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Skin phototype [Number; unit: participants] — Skin phototype definitions according to T.B. Fitzpatrick. This was assessed by the investigator at baseline as:
  II: Always burns easily; tans minimally and with difficulty III:Burns minimally; tans gradually and uniformly (light brown) IV: Burns minimally; always tans well (moderate brown)
  participants
    II | 0 | 1 | 1
    III | 17 | 20 | 37
    IV | 43 | 39 | 82
Atopic Dermatitis (AD) duration [Mean (Standard Deviation); unit: years] | 2.9 (3.4) | 2.7 (2.9) | 2.8 (3.1)
Number of AD acute phase in the last 12 months [Mean (Standard Deviation); unit: episodes] | 4.1 (3.7) | 3.7 (3.3) | 3.9 (3.5)
Duration of the last acute phase [Mean (Standard Deviation); unit: days] | 27.9 (40.8) | 27.0 (53.5) | 27.4 (47.3)
Severity of the last AD acute phase [Count of Participants; unit: Participants]
  Mild | 44 | 41 | 85
  Moderate | 16 | 19 | 35
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — The investigator assessed the global AD severity measurement of erythema and infiltration/papules using IGA on a 6-point scale ranging from 0 = clear (no inflammatory signs of AD) ; 1 = almost clear; 2 = mild disease; 3 = moderate disease, 4 = severe disease; and 5 = very severe disease (severe erythema and severe papulation/infiltration with oozing/crusting), where higher score indicated worst symptoms and decrease in score relates to an improvement in signs and symptoms.
  Participants
    0-Clear | 20 | 22 | 42
    1-Almost clear | 40 | 38 | 78
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: scores on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicated the worse severity of AD.
  scores on a scale
    Erythema | 0.13 (0.21) | 0.10 (0.17) | 0.12 (0.19)
    infiltration / Papulation | 0.09 (0.19) | 0.08 (0.17) | 0.09 (0.18)
    Excoriation | 0.07 (0.15) | 0.10 (0.21) | 0.08 (0.18)
    Lichenification | 0.04 (0.10) | 0.02 (0.07) | 0.03 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse (Quantile 25%)
Description: Time to relapse corresponds to date of relapse - date of baseline. Quantile 25% replaced the median time to relapse that was not reached.
Time Frame: The duration between Baseline and the first AD relapse occurred (up to 89 days)
Population: Analysis was performed on intent-to-treat efficacy (ITT) population that included all participants who were enrolled and randomized.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Moisturizer + Body Wash | Body Wash
Number analyzed (Participants) | 60 | 60
Days | 48 [11 to 86] | 15 [8 to 27]

ADVERSE EVENTS:
Time Frame: 8 months
Description: Analysis was based on safety population that included all treated population.
Arm/Group | Moisturizer + Body Wash | Body Wash
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 14/60 | 17/60
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moisturizer + Body Wash (N=60) | Body Wash (N=60)
PYREXIA (General disorders) | 4 (5) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 6 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. Disclosure agreement covered by contract.